CLINICAL TRIAL: NCT06549153
Title: ACT-Together (Acting on Cancer Testing-Together)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-0236; NCI-2024-06736 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-Together Intervention (Experimental): Participants will be randomized into one of two arms through REDCap
  Interventions: Other: Education Content
- Standard of Care (Experimental): Participants will be randomized into one of two arms through REDCap
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Education Content — Participants will be offered group based education sessions expected to last 90 minutes
  Arms: ACT-Together Intervention
Other: Focus Group — Participants will attend via Zoom
  Arms: Standard of Care

SUMMARY:
To determine the feasibility of a group-based education intervention to improve adherence to recommend surveillance and risk reducing procedures, with a focus at medically underserved women and racial/ethnic minorities with BRCA 1 and 2.

DETAILED DESCRIPTION:
Primary Objective:

To assess the feasibility benchmarks of this intervention by estimating:

1. The enrollment of participants over a 3-month period.
2. Attendance of participants randomized to the ACT-Together Intervention.
3. Completion of baseline and follow up surveys.

Secondary Objectives:

1. Increase breast cancer screening rates or intention to undergo breast cancer screening.
2. Increase uptake of risk-reducing bilateral salpino-oophorectomy (rrBSO) or intention to undergo rrBSO.
3. Demonstrate increase in perceived susceptibility and benefits to risk reducing interventions, and decreased barriers as measured by the Revised Champion Health Belief Scale.

Exploratory Objective:

1. Participant satisfaction with the ACT-Together intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis

   * Arm 1: Diagnosis of MDS intermediate/high/very high risk by Revised International Prognostic Scoring System (IPSS-R), Untreated or up to 2 prior treatments.
   * Arm 2: Diagnosis of relapsed/refractory AML (per European Leukemia Network 2022)[26] receiving treatment as salvage 1-2. MDS or CMML treated with hypomethylating agent (HMA) therapies who progress to AML and have no available better therapies or are not candidates for available therapies, will be eligible at the time of progression to AML.
2. Patients aged ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
4. Temporary prior measures such as apheresis, limited dose cytarabine or use of hydrea while eligibility work-up is being performed are allowed and not counted as a prior salvage
5. In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of protocol therapy will be at least 2 weeks or at least 5 half-lives (whichever is shorter). The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document.
6. The toxicity from prior therapy should have resolved to Grade ≤1, however alopecia and sensory neuropathy Grade ≤2 not constituting a safety risk based on investigators judgement is acceptable.
7. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for patients with controlled CNS leukemia at the discretion of the PI. (2) Use of 1-2 doses of cytarabine (up to 1.5 g/m2 each dose) for patients with rapidly proliferative disease is allowed up to 7 days before the start of study therapy (7 days washout). Use of hydroxyurea for patients with rapidly proliferative disease is allowed on study and before the start of study therapy and will not require a washout. These medications will be recorded in the case-report form.
8. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted. Patients with a known history of CNS disease must have been treated with CNS directed therapy, have at least 2 consecutive LPs with no evidence of CNS leukemia, and must be clinically stable for at least 4 weeks prior to enrollment and have no ongoing neurological symptoms that in the opinion of the treating physician are related to the CNS disease

Serum biochemical values with the following limits:

1. Patients must have adequate renal function as demonstrated by a creatinine clearance (CrCl) ≥ 40 mL/min calculated by either the Cockcroft-Gault formula, Modification of Diet in Renal Disease (MDRD) eGFR or measured by 24 hours' urine collection. For patients with BMI >23, Adjusted body weight and not Ideal Body Weight is the recommended parameter.
2. Direct bilirubin <1.5 x ULN unless considered due to Gilbert's syndrome
3. Aspartate aminotransferase or alanine aminotransferase ≤2.0 x ULN (aspartate aminotransferase or alanine aminotransferase ≤3.0 x ULN if deemed related to leukemia by the treating physician) 10. White blood cell count <10 x 109/L. Hydroxyurea may be used to reduce the WBC count to < 10x109/L.

   11. Ability to understand and provide signed informed consent. 12. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment 13. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 4 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.

   Exclusion Criteria:

   Patients with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which could compromise participation in the study.

   2. Patients on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed.

   3. Prior organ transplantation including allogenic stem-cell transplantation within 3 months prior to planned enrollment, active graft versus host disease (GVHD) >Grade 1 or requiring transplant-related immunosuppression with the exception of low dose cyclosporine and tacrolimus.

   4. Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia.

   5. Patients with a known HIV infection that is not well controlled (i.e. any detectable circulating viral load) at the time of enrollment.

   6. Patients with known positive hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months (Hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.

   7. Patients who have had any major surgical procedure within 14 days of Day 1. 8. Other severe acute or chronic medical conditions that is active and not well controlled including colitis, inflammatory bowel disease, or psychiatric conditions including active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

   9. Active and uncontrolled disease (active infection requiring systemic therapy or fever likely secondary to infection within prior 48 hours): prophylactic antibiotics or prolonged course of IV antibiotics for controlled infection are allowed, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure NYHA class III/IV, clinically significant and uncontrolled arrhythmia, as judged by the treating physician.

   10. Requirement to use anti-TNF drugs (infliximab, etanercept, adalimumab, certolizumab, golimumab).

   11. Patients unwilling or unable to comply with the protocol. 12. Live vaccination within 28 days from start of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jose Rauh-Hain, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org